CLINICAL TRIAL: NCT07072143
Title: The PARTNER Study - An International Prospective Observational Study on Pediatric Patients With Very Rare Tumors.
Brief Title: An International Study on Pediatric Patients With Rare Tumors.
Acronym: PARTNER
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliera di Padova (Other)
Collaborators: St. Anna Children's Hospital, Vienna (Unknown); Children's Hospital Zagreb (Other); Centre Hospitalier Universitaire de La Réunion, FRANCE (Unknown); Klinikum Dortmund (Unknown); University Children's Hospital Tuebingen (Other); Hellenic Oncology Research Group (Other); Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other); Kaplan Medical Center, Rehovot, Israel (Unknown); Vilnius University hospital Santaros klinikos, Vilnius, Lithuania (Unknown); University of Skopje (Other); Gdansk Medical University (Poland) (Unknown); Centro Hospitalar do Porto (Other); Bucharest Emergency Hospital (Other); Institute for Oncology and Radiology Serbia, Belgrade (Unknown); University Hospital Bratislava (Other); University Medical Centre Ljubljana (Other); University of Bilbao (Unknown); Göteborg University (Other); University Hospital, Paris (Other)
Responsible Party: Principal Investigator, Gianni Bisogno, Professor of Paediatrics, Azienda Ospedaliera di Padova
Other Study IDs: The PARTNER study (AOP3417)
Record Dates: First submitted 2025-04-15; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Paraganglioma/ Phaeochromocytoma; Melanoma and Other Malignant Neoplasms of Skin; Gastrointestinal Stromal Tumor (GIST); Adrenocortical Tumor; Pancreatic Tumors; Esthesioneuroblastoma, Olfactory; Mesothelioma; Nasopharyngeal Carcinoma (NPC); NUT Carcinoma; Pleuropulmonary Blastoma; Salivary Gland Tumors; Thymic Tumors; Thyroid Carcinoma; Appendiceal Cancers
Keywords: children; rare tumors; very rare tumors; adolescents; PARTNER Study
MeSH Terms: conditions — Melanoma; Gastrointestinal Stromal Tumors; Adrenal Cortex Neoplasms; Pancreatic Neoplasms; Esthesioneuroblastoma, Olfactory; Mesothelioma; Nasopharyngeal Carcinoma; Pleuropulmonary blastoma; Thymus Neoplasms; Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The PARTNER study is an international, prospective, observational study of paediatric patients with very rare tumours.

DETAILED DESCRIPTION:
There are some very rare tumors (with an annual incidence of less than two per million children) that can affect children and adolescents. These neoplasms include a wide variety of cancers; some are rare at any age, while others are typical of adults but very rare in children. Due to their rarity, studies have so far been scarce, often lacking univocal diagnostic criteria, and more information is needed to improve treatment outcomes.

The aim of this study is to collect epidemiological, clinical, biological, radiological and treatment data on children and adolescents with rare cancers in order to improve our understanding of these tumors and how their clinical and biological characteristics affect treatment outcomes.

Due to the rarity of these malignancies, international collaboration is necessary to collect sufficient data on each tumour type.

While the investigators are not proposing specific treatments, the data collected will inform recommendations for the diagnosis and treatment of patients.

The PARTNER Study is an observational, prospective study. It is sponsored by Padua University Hospital AOUP (Italy), and all European centres collaborating with the EXPeRT group have been invited to participate. It is a non-profit study, meaning it has no commercial purpose, only the aim of improving knowledge and treatment for children with rare cancers. PARTNER activities are supported in different countries by national funds, as well as by the European Commission through the European Reference Network for Paediatric Oncology (ERN PaedCan). Please visit https://paedcan.ern-net.eu/ for more information.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents (age 0-18 years) with a primary or relapsed Very Rare Tumor diagnosed and/or treated in a participating country/center.
* Written informed consent from the patient and/or the parent/legal guardian

Exclusion Criteria:

* Absence of Written informed consent from the patient and/or the parent/legal guardian

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents (0-18 years) with a primary or relapsed Very Rare Tumor (VRT)
Sampling Method: Non-Probability Sample
Enrollment: 6250 (Estimated)
Dates: Start 2025-01-25 (Actual); Primary Completion 2049-01-06 (Estimated); Study Completion 2049-06-06 (Estimated)

PRIMARY OUTCOMES:
Epidemiology | through study completion, an average of 1 year
  Evaluate the number of patients (aged 0-18 years) with different Very Rare Tumors in the different countries: observed cases will be compared with expected cases.
Use of International Recommendations | through study completion, an average of 1 year
  The study aims to measure the number of patients treated for different neoplasms in different countries, and the proportion of those treated in accordance with the International Recommendations.
Survival of children and adolescents (0-18 years) affected by Very Rare Tumors | through study completion, an average of 1 year
  The study will correlate the clinical characteristics of the tumor (size, site, extension) with the treatment, the risk of recurrence and survival.

CONTACTS AND LOCATIONS:
Overall Officials: Gianni Bisogno, MD, Principal Investigator — Azienda Ospedale Università Padova - Italy
Locations (1):
- Pediatric Oncology Unit, University Hospital Padova [AOUP Azienda Ospedale Università Padova], Padua, Italy, Italy

REFERENCES:
- [Background] Orbach D, Ferrari A, Schneider DT, Reguerre Y, Godzinski J, Bien E, Stachowicz-Stencel T, Surun A, Almaraz RL, Dragomir M, Jani D, Ami TB, Roganovic J, Brecht IB, Ladenstein R, Bisogno G. The European Paediatric Rare Tumours Network - European Registry (PARTNER) project for very rare tumors in children. Pediatr Blood Cancer. 2021 Jun;68 Suppl 4:e29072. doi: 10.1002/pbc.29072. Epub 2021 Apr 29. PMID 33913610
- See also: The page describes the PARTNER project inside the website of SIOP Europe (the European Society for Paediatric Oncology) — https://www.raretumors-children.eu/partner-project/